CLINICAL TRIAL: NCT06692621
Title: Effects of Carbetocin and Oxytocin Used in Cesarean Sections on Postoperative Pain
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Other Study IDs: E2-234595
Record Dates: First submitted 2024-10-21; First posted 2024-11-18 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: PREG1
Keywords: carbetocin; oxytocin; cesarean analgesia
MeSH Terms: interventions — Oxytocin; carbetocin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- O:oxytocin: In the oxytocin group, oxytocin ('Synpitan forte 5 IU/ml im/iv ampoule, Deva İlaç Sanayi, Turkey)' was administered 20 IU intravenously (5 IU intravenous bolus followed by 15 IU/hour infusion) in accordance with the recommendations of the Ministry of Health of the Republic of Turkey.
  Interventions: Drug: Oxytocin
- C:carbetocin: In the carbetocin group, carbetocin 'Pabal 100 microgram/ml iv solution for injection ampoule, Ferring GmbH, Germany) was diluted with 20 ml of 0.9% NaCl solution and administered over 30-60 seconds.
  Interventions: Drug: Carbetocin

INTERVENTIONS:
Drug: Oxytocin — Medicines were administered in appropriate doses
  Other Names: Deva İlaç Sanayi, Turkey
  Groups: O:oxytocin
Drug: Carbetocin — Medicines were administered in appropriate doses
  Other Names: Ferring GmbH, Germany
  Groups: C:carbetocin

SUMMARY:
The aim of this observational study is to compare postoperative analgesic consumption in patients who received peroperative carbetocin or oxytocin. The main question it aims to answer is:

. Does peroperative carbetocin use reduce postoperative analgesic consumption compared to oxytocin?

Patients who receive routine uterotonic agents in caesarean section surgeries will be divided into two groups and their postoperative 24-hour analgesic consumption will be compared.

DETAILED DESCRIPTION:
Postpartum hemorrhage (PPH) is one of the most important causes of perioperative maternal deaths. Oxytocin and carbetocin are the most important uterotonic agents used for PPH. Oxytocin has a half-life of 4-10 minutes (min) and can provide continuous uterotonic properties through infusion. Carbetocin, which has been used increasingly in recent years, is a synthetic analogue of oxytocin and has a strong uterotonic effect on oxytocin receptors. Oxytocin, which is used in PPH prophylaxis and management in cesarean delivery, has some maternal side effects depending on the rate of administration. These are cardiovascular effects, nausea, vomiting, headache and allergic reactions. Since it is structurally similar to vasopressin, water retention in the body and hyponatremia, convulsions and coma can be seen, although rarely. The most common cardiac effects after oxytocin administration are dose-dependent hypotension and tachycardia. Smooth muscle relaxation caused by stimulation of calcium-dependent nitrite oxide is held responsible for hypotension.[3] Carbetocin, a long-acting oxytocin analog, has similar side effects and further research is needed on its effectiveness.

There are potential studies supporting that the oxytocinergic system affects pain perception. Oxytocin released into the central nervous system plays an important role in the transmission and modulation of pain signals. Glutamatergic activation of oxytocin in the dorsal root ganglia results in GABAergic inhibition of Aδ and C fibers that play a role in nociception. Carbetocin is also thought to have similar effects in analgesia. Although there are studies showing that carbetocin reduces postoperative analgesic use compared to oxytocin , there is no clear consensus in the literature on this subject. The studies conducted by De Bonis et al. and Gawecka et al. were guiding in designing this study. While De Bonis et al. found that carbetocin reduces analgesic consumption, Gawecka et al. could not show a significant difference between the two agents.

In this study, the investigators aim to contribute to the literature by comparing the analgesic activities of oxytocin and carbetocin to observe the differences in hemodynamic and other side effects of these two agents.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in the American Society of Anesthesiologists (ASA) II class,
* who have had a previous uncomplicated cesarean delivery,
* who are 18-45 years old and are planned to undergo elective cesarean section with spinal anesthesia technique

Exclusion Criteria:

* Patients who cannot use the patient controlled analgesia (PCA) device postoperatively,
* have limited intellectual function
* have contraindications for spinal anesthesia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only pregnant women were included in our study.
Study Population: Pregnant women between the ages of 18-45
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2024-10-04 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Postoperative 24-hour analgesic consumption (Total tramadol mg / 24 hours ) | 04/10/2024-04/01/2025
  analgesic consumption

SECONDARY OUTCOMES:
amount of intraoperative bleeding (Preoperative / postoperative hemoglobin g/dl ) | 04/10/2024-04/01/2025
  intraoperative bleeding
Postoperative 24-hour Heart rate variables (/minute) | 04/10/2024-04/01/2025
  Postoperative 24-hour hemodynamic variables
Postoperative 24-hour arterial blood pressure variables (mmHg) | 04/10/2024-04/01/2025
  Postoperative 24-hour hemodynamic variables
Postoperative 24-hour oxygen saturation variables (%) | 04/10/2024-04/01/2025
  Postoperative 24-hour hemodynamic variables

CONTACTS AND LOCATIONS:
Overall Officials: Havva Esra Türkyılmaz Uyar, Study Director — esrauyarturkyilmaz@yahoo.com
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Bonis M, Torricelli M, Leoni L, Berti P, Ciani V, Puzzutiello R, Severi FM, Petraglia F. Carbetocin versus oxytocin after caesarean section: similar efficacy but reduced pain perception in women with high risk of postpartum haemorrhage. J Matern Fetal Neonatal Med. 2012 Jun;25(6):732-5. doi: 10.3109/14767058.2011.587920. Epub 2011 Jul 15. PMID 21761999
- [Background] Gawecka E, Rosseland LA. A secondary analysis of a randomized placebo-controlled trial comparing the analgesic effects of oxytocin with carbetocin: postcesarean delivery morphine equivalents. Anesth Analg. 2014 Oct;119(4):1004. doi: 10.1213/ANE.0000000000000372. No abstract available. PMID 25232698
- See also: main source — https://pubmed.ncbi.nlm.nih.gov/21761999/
- See also: main source — https://pubmed.ncbi.nlm.nih.gov/25232698/
- Available data/document: Individual Participant Data Set: Yöktez — https://tez.yok.gov.tr/UlusalTezMerkezi/tezlerim.jsp?sira=0 — You can reach us at harunzengin71@gmail.com